CLINICAL TRIAL: NCT04879524
Title: Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis for the Treatment of Dyssynergic Defaecation: a Prospective Observational Study
Brief Title: Infracoccygeal Botox for Dyssynergia
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 291709
Record Dates: First submitted 2021-04-28; First posted 2021-05-10 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dyssynergic Defaecation; Evacuation Disorder; Anismus; Defecation Disorder
Keywords: Botulinum toxin type A; Botox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous infracoccygeal Botulinum toxin injection to puborectalis: 100 units of Botulinum toxin type A (Botox, Allergan, Ireland) injection into the puborectalis muscle to each side of the midline, achieving a total of 200 units
  Interventions: Procedure: Percutaneous infracoccygeal Botulinum toxin injection to puborectalis

INTERVENTIONS:
Procedure: Percutaneous infracoccygeal Botulinum toxin injection to puborectalis — The intervention is an injection of 200 units of Botulinum toxin type A in to the puborectalis muscle under ultrasound guidance.
  In the prone position, the puborectalis muscle will be identified below the coccyx using ultrasound. After skin preparation using 70% Isopropyl Alcohol Pad, and up to 5ml of local anaesthetic (1% lidocaine), an electromyography (EMG) needle will be inserted and the puborectalis muscle stimulated using a current to confirm correct needle position. 200 units of BTXA (Botox, Allergan, Ireland) prepared in 2 ml of saline solution and drawn up using a 2ml syringe. 1ml (100 units) of BTXA solution is injected through the EMG needle into the puborectalis muscle to each side of the midline, achieving a total of 200 units. The needle is withdrawn, and the procedure is complete.

SUMMARY:
Background:

Constipation is a common problem, affecting up to 20% of the population during their lifetime. Some patients respond poorly to standard treatments such as laxatives. A subgroup of these have dyssynergic defaecation where the muscles that control bowel movements fail to relax during pushing, preventing evacuation of stools. Currently, the mainstay of treatment requires muscle retraining by a therapist using a technique called biofeedback. Patients in whom biofeedback has failed are left with few options, one of which includes Botox injection into the pelvic floor muscles involved in the defaecation process. However, current method of injection is inaccurate and often requires anaesthesia. The investigators propose a novel technique for Botox delivery which reduces the risks and associated costs.

Objectives:

1. The primary objective is to demonstrate technical feasibility of percutaneous infracoccygeal Botox injection as an alternative to transanal puborectalis muscle injection for the treatment of dyssynergic defaecation.
2. The secondary objectives are to assess the safety and acceptability of this technique, and to derive pilot clinical effectiveness data to inform future studies.

Methods:

The investigators will carry out Botox injection into the puborectalis muscle under ultrasound guidance in the outpatient department. This will be done by percutaneous injection below the coccyx where the puborectalis has been demonstrated to be easily accessible. An electromyography of the puborectalis is obtained before the injection to demonstrate proof of mechanism. The investigators will collect data using a combination of questionnaires, patient baseline data, and anorectal physiology test results before and after the treatment.

Outcomes:

* Feasibility: procedure duration, rate of identification of puborectalis by ultrasound scan and pre-injection EMG, procedure limitations, and successful injection rate
* Safety: rate of adverse events
* Acceptability: patient pain and comfort, willingness to undergo repeat procedure
* Preliminary data on effectiveness: Cleveland Clinic constipation score, anorectal physiology test results

DETAILED DESCRIPTION:
Patients with dyssynergic defaecation represent a subgroup of a larger group of patients presenting with symptoms of chronic constipation. The disorder is characterised by impaired stool expulsion as a result of inappropriate contraction of the pelvic floor musculation despite normal propulsive force during attempted defaecation. Failure of the puborectalis and/or anal sphincter muscles to relax during evacuation leads to a closed anal canal which prevents the emptying of stools.

A Cochrane review in 2014 on the treatment of chronic constipation in adults demonstrated a high prevalence of dyssynergic defaecation and a variety of treatments. In this group, biofeedback was found to be superior to oral diazepam, sham treatment, and laxatives; while surgical procedures such as partial division of the puborectalis muscle were more efficacious, the risks of adverse reaction, namely incontinence, were high. Thus, biofeedback therapy is the current gold-standard for the treatment of dyssynergia. The success rate of biofeedback in correcting or improving the symptoms in patients with dyssynergia varies between 33% and 80%. Difficulty arises in those in whom biofeedback is unsuccessful, as there is little, and conflicting, low quality evidence on alternative therapies.

One further therapeutic option uses injection of Botulinum toxin type A (BTXA) into the puborectalis and/or external anal sphincter muscles. This is currently the second-line treatment for dyssynergic defaecation in whom biofeedback has failed. A systematic review in 2016 on the use of BTXA in patients with 'anismus', a term previously used to describe dyssynergic defaecation, demonstrated initial clinical improvement in symptoms in 77.4% of patients. Two of the seven studies were conducted on participants in whom biofeedback therapy had failed. Complications were reported in 7.4% of patients (0 to 22.6%) and included faecal incontinence, which was minor and transient, posterior anal fissure, and rectal prolapse. The effect of BTXA was not permanent, with clinical improvement declining to 46% at four months after the injection. For this reason, several studies offered repeated treatments.

The delivery of BTXA injection varied between studies and institutions in terms of dosage and position of injection, but all were performed via perianal or transanal approaches, often requiring sedation or anaesthesia. There are several disadvantages of this approach including cost (operating theatre utilisation) and risks associated with anaesthesia and infection from passing the needle through a contaminated operative field. In addition, the injection site is defined blind by the surgeon's finger (an issue of accuracy of injection and hazard of needle stick injury).

The proposed study aims to demonstrate the technical feasibility of an alternative approach to delivering BTXA injection in adult patients with dyssynergic defaecation. This novel technique injects BTXA into the puborectalis muscle percutaneously using an infracoccygeal approach under ultrasound guidance. This allows the procedure to be performed in an outpatient radiology setting without the need for any form of anaesthesia or analgesia. The injection is performed in a clean operative field away from the anus, minimising risk of infection and the muscle can be clearly visualised (see below). These advantages will be particularly valuable in patients who require repeated procedures or those with multiple co-morbidities at high anaesthetic risk.

The utilisation of BTXA in human is well established. This medication is licensed for use in focal spasticity with well-established side-effects and interactions. Current evidence for the use of BTXA in dyssynergic defaecation is based on the conventional transanal approach, with report on efficacy and complications as previously stated.

The puborectalis is easily accessible below the coccyx, and is the site for ultrasonic assessment in the paediatric population. The identification of puborectalis muscle in the infracoccygeal position has not been described in the literature in the adult population. However, pilot imaging studies on a small number of non-obese subjects have been successful in easily identifying the puborectalis using ultrasound scan. This approach has the potential to allow accurate administration of BTXA injection under ultrasonic guidance in the outpatient setting without the need for anaesthesia or operating theatre utilisation. The general aim of this study is to demonstrate that percutaneous infracoccygeal BTXA injection is a valid alternative approach to transanal injection for the treatment of dyssynergic defaecation. Specifically, the investigators will determine technical feasibility (including pilot proof of mechanism), patient acceptability, safety, and pilot efficacy outcomes for a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 80 years
* Diagnosis of dyssynergic defaecation using Rome IV criteria
* Ability to understand written and spoken English
* Ability and willingness to give informed consent

Exclusion Criteria:

* Paediatric patients (age under 18 years)
* Diagnosis of defined structural or metabolic diseases that could cause constipation, such as Hirschsprung's disease, Parkinson's disease, multiple sclerosis, hypothyroidism (untreated), diabetic neuropathy, muscular dystrophy, motor neurone diseases, spinal injury leading to paraplegia, cauda equina syndrome
* Psychiatric or physical inability to comply with the study protocol (including e-diary assessments) at investigator discretion.
* Contra-indications to BTXA such as allergies, pregnancy (or intention to become pregnant during study period), breastfeeding, generalised disorders of muscle activity, myasthenia gravis
* Contra-indications to infracoccygeal injection at injection site such as infection or pressure sore, spina bifida, pilonidal disease, bleeding disorders (including therapeutic anticoagulation)
* Morbid obesity (BMI ≥ 40)
* Defunctioning loop or end stoma in situ
* External rectal prolapse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with dyssynergic defaecation using Rome IV criteria
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Knowles, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis: 100 units of Botulinum toxin type A (Botox, Allergan, Ireland) injection into the puborectalis muscle to each side of the midline, achieving a total of 200 units
  Percutaneous infracoccygeal Botulinum toxin injection to puborectalis: The intervention is an injection of 200 units of Botulinum toxin type A in to the puborectalis muscle under ultrasound guidance.
  In the prone position, the puborectalis muscle will be identified below the coccyx using ultrasound. After skin preparation using 70% Isopropyl Alcohol Pad, and up to 5ml of local anaesthetic (1% lidocaine), an electromyography (EMG) needle will be inserted and the puborectalis muscle stimulated using a current to confirm correct needle position. 200 units of BTXA (Botox, Allergan, Ireland) prepared in 2 ml of saline solution and drawn up using a 2ml syringe. 1ml (100 units) of BTXA solution is injected through the EMG needle into the puborectalis muscle to each side of the midline, achieving a total of 200 units. The needle is withdrawn, and the procedure is complete.
Period: Overall Study
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Started | 8
Completed | 6
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Identification of Puborectalis During Ultrasound Scan
Description: The investigator will record the number of times the puborectalis muscle is successfully identified using ultrasound scan (muscle seen to contract on volition) and pre-injection EMG (change in EMG waveform on volitional contraction) by the radiologist and neurologist, respectively, at the beginning of the injection procedure.
Time Frame: Visit 3: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Procedure Duration
Description: The investigator will record the time (in minutes) taken to for the radiologist to complete the injection procedure
Time Frame: Visit 3: week 18
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
minutes | 5 [5 to 10]

3. Primary Outcome: Procedure Limitations
Description: The investigator will record any procedure or patient related factors which prevented a successful injection, e.g. body habitus or equipment failure.
Time Frame: Visit 3: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Rate of Adverse Events
Description: Any adverse events reported by the patients or their clinician following the injection
Time Frame: From visit 3 to visit 6: week 18 to 42
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Participants | 0

5. Secondary Outcome: Patient's Level Pain and Comfort Assessed at Post-procedure
Description: Following the procedure, the patient will complete a post-procedure questionnaire.
  * The patient is asked to give their response to the statement "the procedure was painful" on a 5-point rating scale (strongly agree/ agree/ neutral/ disagree/ strongly disagree).
  * The patient is asked to give their response to the statement "the procedure was comfortable" on a 5-point rating scale (strongly agree/ agree/ neutral/ disagree/ strongly disagree).
Time Frame: Visit 3: week 18
Population: Reported pain
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Participants | 2

6. Secondary Outcome: The Number of Patient Indicating *Yes*, They Would be Willing to Undergo a Repeat Procedure
Description: The number of patients who answered Yes when asked if they will be willing to undergo a repeat procedure (yes/no) in a post-procedure questionnaire.
Time Frame: Visit 3: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Percutaneous Infracoccygeal Botulinum Toxin Injection to Puborectalis
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04879524/Prot_SAP_000.pdf